CLINICAL TRIAL: NCT06272201
Title: Incisionless Suture Plications in a POSE2.0 Interventional Randomized Obesity Study (The INSPIRO Study)
Brief Title: Incisionless Suture Plications in a POSE2.0 Interventional Randomized Obesity Study
Acronym: INSPIRO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: USGI Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50620 TPR
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): POSE2.0 Treatment with Lifestyle Modification
  Interventions: Device: POSE2.0 procedure with g-Cath EZ Delivery Catheter with Snowshoe Suture Anchors
- Control (No Intervention): Lifestyle Modification alone

INTERVENTIONS:
Device: POSE2.0 procedure with g-Cath EZ Delivery Catheter with Snowshoe Suture Anchors — POSE2.0 (g-Cath EZ snowshoe suture anchors placed in the mid + distal body without placement in the fundus), with a moderate intensity diet and exercise program
  Arms: Treatment

SUMMARY:
This is a multi-center, open-label, 2-group randomized pivotal study evaluating a minimally invasive weight loss procedure. The intent is to evaluate the safety and effectiveness of POSE2.0 (sutures placed in the mid + distal body without placement in the fundus), with a moderate intensity diet and exercise program, as compared to diet and exercise alone. The procedure will be performed using the g-Cath EZ Delivery Catheter with Snowshoe Suture Anchors (AKA g-Cath or g-Cath EZ) and associated devices (g-Prox EZ, g-Lix and Transport), known collectively as the Incisionless Operating Platform (IOP).

DETAILED DESCRIPTION:
This is a multi-center, open-label, 2-group randomized pivotal study evaluating a minimally invasive weight loss procedure. The intent is to evaluate the safety and effectiveness of POSE2.0 (g-Cath EZ Snowshoe Suture Anchors placed in the mid + distal body without placement in the fundus), with a moderate intensity diet and exercise program, as compared to diet and exercise alone. The procedure will be performed using the g-Cath EZ Delivery Catheter with Snowshoe Suture Anchors (AKA g-Cath or g-Cath EZ) and associated devices (g-Prox EZ, g-Lix and Transport), known collectively as the Incisionless Operating Platform (IOP).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Subject agrees to be compliant with study requirements and adhere to post-operative dietary & exercise recommendations for the duration of the study.
3. Subjects between the ages of 22-65 years.
4. History or failure with non-surgical weight-loss methods.
5. If female, be either post-menopausal, surgically sterile, or agree to practice birth control during year of study and have negative serum HCG at screening/baseline.
6. Have a Body Mass Index (BMI) of ≥ 30 and ≤ 50 kg/m².
7. Absence of current severe systemic disease (including, but not limited to: coronary artery disease, chronic obstructive pulmonary disease, congestive heart failure, cancer, and chronic renal disease).
8. Agrees to forego any additional weight loss interventional procedures or liposuction for 12 months following study enrollment.
9. Have not taken any prescription or over-the-counter weight loss medications in the last 6 months, with exception of medications used to manage T2D so long as the subject has been on a stable dose and weight has persisted.
10. Residing within a reasonable distance from the Investigator's treating office (~50 miles) and willing and able to travel to the Investigator's office to complete all routine follow-up visits.

Exclusion Criteria:

1. History of or intra-operative evidence of prior bariatric, gastric or esophageal surgery.
2. Esophageal stricture or other anatomy and/or condition that could preclude passage of endoluminal instruments or procedure execution.
3. Moderate gastro-esophageal reflux disease (GERD), defined as symptoms that cause subject severe discomfort, compromise performance of daily activities, and/or condition is not entirely controlled with drug therapy.
4. Large hiatal hernia (>3 cm) by history or as determined by pre-enrollment endoscopy.
5. Pancreatic insufficiency/disease.
6. History of gastroparesis or symptoms that would be suggestive of gastroparesis or generalized dysmotility (e.g., esophago-gastric motility issues and lower esophageal sphincter abnormalities).
7. Patients who are known to be pregnant or breast-feeding, or plan to become pregnant in the next 12 months.
8. History of a known diagnosis or pre-existing symptom of rheumatoid arthritis, scleroderma, system lupus, or other autoimmune connective tissue disorder.
9. Immunosuppressive medications or systemic steroids (i.e., oral prednisone) within 6 months of Visit 1. Intranasal/inhaled steroids are acceptable.
10. Unable or unwilling to avoid use of aspirin and/or non-steroidal anti-inflammatory drugs (NSAIDs), or other medications known to be gastric irritants beginning two weeks prior to enrollment and throughout the entire study.
11. History of inflammatory disease of the GI tract; coagulation disorders; hepatic insufficiency or cirrhosis.
12. Active gastric erosion, lesion, or gastric/duodenal ulcer.
13. History of or current platelet or coagulation dysfunction, such as hemophilia.
14. History or present use of insulin or insulin derivatives for treatment of diabetes.
15. Patients with type II diabetes mellitus on oral agents (not injectables) with HgA1c > 9 at the time of enrollment.
16. Active smoker or someone who has been a smoker in the 6 months leading up to the study.
17. Portal hypertension and/or varices.
18. Patient has a history of drug or alcohol abuse or positive at screening for drug use.
19. Patient is currently using marijuana/cannabis for either medicinal or recreational use, or has plans to start using over the next 12 months.
20. Present or history of psychosis, bipolar disease, obsessive-compulsive disorder, binge eating, and/or other eating disorders after pre-enrollment history and medical /psychological assessment.
21. Beck Depression Inventory (Short) Score ≥ 12, and/or uncontrolled depression after pre-enrollment psychological and medical assessment.
22. Patient score >2 in any of the identified symptoms in the nausea/vomiting or bloating/distension domains on the Gastroparesis Cardinal Symptom Index (GCSI).
23. Non-ambulatory or has significant impairment of mobility (i.e. cannot ambulate for 30 minutes).
24. Known hormonal or genetic cause for obesity including untreated hypothyroidism (TSH >5.0 U/ml).
25. Present or history of chronic abdominal pain.
26. Participating in another clinical study that could compromise compliance with the POSE2.0 study (must be cleared with investigator and USGI Medical).
27. Subjects with a personal history of allergic/anaphylactic reactions including hypersensitivity to the drugs or materials that will be utilized in the study procedure.
28. Any other medical condition that would not permit elective endoscopy such as poor general health or history and/or symptoms of severe renal, hepatic, cardiac, and/or pulmonary disease, and/or physician's assessment that the subject is not an appropriate candidate.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of total body weight loss (%TBWL) following randomization | 12 months
  To be deemed effective, the difference in %TBWL between the treatment group minus the control group must be significantly greater than 5%.
Responder rate of at least 50% in the POSE2.0 treatment group | 12 months
  Responder defined as >5% TBWL
Safety- Incidence of device and procedure related adverse events through 12 months | 12 months
  Incidence of device and procedure related adverse events through 12 months defined as Clavien-Dindo Class III or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Barham Abu Dayyeh, MD, MPH, Principal Investigator — Mayo Clinic; Erik Wilson, MD, Principal Investigator — University of Texas Medical School at Houston

IPD SHARING:
Plan to Share IPD: No